CLINICAL TRIAL: NCT02487082
Title: Pilot Study of Sleep Therapy and Biomarkers in Children With Autism Spectrum Disorders
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: too few subjects enrolled
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Jill Miller-Horn, Assistant Professor of Neurology and Pediatrics, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 65708
Record Dates: First submitted 2015-06-29; First posted 2015-07-01 (Estimated); Results first posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-05

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; Children; Melatonin; Donepezil; Sleep disorder
MeSH Terms: conditions — Autism Spectrum Disorder; Sleep Wake Disorders | interventions — Melatonin; Donepezil

STUDY DESIGN:
Intervention Model Description: The study is conducted in 2 main phases, supplemented by an initial Run-In Phase and a Final Wash-Out Phase.
  The Run-In phase (5 weeks) - All subjects receive Placebo and instructions about how to improve sleep hygiene. This allows us to evaluate a) response to placebo and b) the effect of improved sleep hygiene in the absence of study drug in both groups.
  Phase 1 (5 weeks) - Group A receives study drug (donepezil & melatonin). Group B receives Placebo. Here we assess the benefit of study drug vs. Placebo in a parallel group design.
  Phase 2 (5 weeks) - Both groups receive study drug (donepezil & melatonin). Here we assess the effect of switching from Placebo to study drug in Group B, and the effect of an extra 5 weeks of study drug in Group A.
  Wash-Out Phase (variable length, 2-12 weeks) - study drug is discontinued.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (Other): Run-In Phase: Placebo. Phase 1 & Phase 2: Melatonin and donepezil (melatonin 3mg and donepezil 1.25-5mg based on age/weight each night) for 10 weeks Wash-Out Phase: no active or placebo medication. Note: Dosage of study drug varies with age/weight. Younger children (<12 years or < 80 lbs. weight start at a lower dose of donepezil (1.25 mg/night) and increase to 2.5 mg/night after one week. Older children (>= 12 years or >= 80 lbs weight) start at 3 mg donepezil and increase to 5 mg after one week. The dose of melatonin remains stable at 3 mg throughout for both groups.
  Interventions: Drug: Melatonin and Donepezil; Other: Placebo
- Group B (Other): Run-In Phase: Placebo. Phase 1: Placebo. Phase 2: Melatonin and donepezil (melatonin 3mg and donepezil 1.25-5mg based on age/weight each night) or placebo for 5 weeks Wash-out Phase: no active or placebo medication. Note: Dosage of study drug varies with age/weight. Younger children (<12 years or < 80 lbs. weight start at a lower dose of donepezil (1.25 mg/night) and increase to 2.5 mg/night after one week. Older children (>= 12 years or >= 80 lbs weight) start at 3 mg donepezil and increase to 5 mg after one week. The dose of melatonin remains stable at 3 mg throughout for both groups.
  Interventions: Drug: Melatonin and Donepezil; Other: Placebo

INTERVENTIONS:
Drug: Melatonin and Donepezil — 10 weeks of active study medication in Group A during Phase 1 & Phase 2. 5 weeks of active study medication in Group B during Phase 2.
  Other Names: Aricept
Other: Placebo — For both groups: 5 weeks of Placebo in the Run-In Phase. For Group B: an addition 5 weeks of Placebo in Phase 1.

SUMMARY:
The purpose of this study is to test the combined effect of melatonin and donepezil on improving sleep and behavior in children with Autism Spectrum Disorders. Melatonin is a natural neurohormone that helps regulate sleep and wake cycles. Donepezil is used to improve mental function for people with Alzheimer's disease. Children with Autism Spectrum Disorders are more likely to have problems sleeping than other children. This difficulty has been linked to daytime behavioral problems and family stress.

DETAILED DESCRIPTION:
The goal of the present exploratory investigation is to see if there is a suggestion of a large additive or synergistic effect of melatonin and donepezil given together. Individually both medications improve sleep, but appear do so in different ways, with melatonin altering circadian rhythm and donepezil altering the characteristics of REM sleep. In this pilot investigation we will examine whether their combined effects on sleep lead to a large improvement in the behavior of children with ASD. Combined pharmacotherapy is very common in clinical practice, but is rarely studied in research (Comer et al. 2010). These two medications are both well tolerated and there is no negative drug interaction between the two. This investigation will use an RCT as well as a set of exploratory analyses to assess the combined effects of these two medications compared to placebo in terms of behavioral and sleep measures. In addition we will collect exploratory biomarkers (e.g., digit ratio, the ratio of the lengths different fingers as a measure of the balance of sex hormones during embryonic development) to relate to the various sleep and behavioral measures. A positive signal from this study may be used to guide a follow-up study with greater numbers of study subjects and statistical power.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female children
* Ages 4 to 17 1/2 years
* Diagnosis with Autism Spectrum Disorder on the basis of the clinical judgment of an autism specialist, preferably using the Autism Diagnostic Observation Schedule or the Autism Diagnostic Interview-Revised.

Exclusion Criteria:

* Abnormal electroencephalogram in the past month
* Cardiovascular problems
* Asthma
* Respiratory disease
* Peptic ulcer disease
* Renal or hepatic dysfunction (abnormal blood urea nitrogen/creatinine or 2 times elevated liver transaminases)
* Urinary tract obstruction
* Underweight (body mass index < 5th percentile compared to age and sex matched population)
* Other serious illness
* Use of any of the following drugs that might interact with study medications (anticholinergics, systemic corticosteroids, phenobarbital, peginterferon, beta-blockers or any drug that may cause arrhythmias). Drugs that induce or inhibit cytochrome P450 2D6 and cytochrome P450 3A4 (enzymes important for drug metabolism) will be allowed because any effects of such medications are likely to be lost in individual variability due to genetic polymorphisms.
* Use of medications affecting sleep with a half-life of 7 days or more. [Children on medications affecting sleep with a half-life of less than 7 days (including melatonin and donepezil) are eligible if they agree to discontinue use for the duration of the trial.]
* Pregnancy and lactation

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2015-06; Primary Completion 2020-12-31 (Actual); Study Completion 2021-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill Miller-Horn, MD, MS, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook University, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buckley AW, Sassower K, Rodriguez AJ, Jennison K, Wingert K, Buckley J, Thurm A, Sato S, Swedo S. An open label trial of donepezil for enhancement of rapid eye movement sleep in young children with autism spectrum disorders. J Child Adolesc Psychopharmacol. 2011 Aug;21(4):353-7. doi: 10.1089/cap.2010.0121. PMID 21851192
- [Background] Cidav Z, Marcus SC, Mandell DS. Implications of childhood autism for parental employment and earnings. Pediatrics. 2012 Apr;129(4):617-23. doi: 10.1542/peds.2011-2700. Epub 2012 Mar 19. PMID 22430453
- [Background] Malow BA, Marzec ML, McGrew SG, Wang L, Henderson LM, Stone WL. Characterizing sleep in children with autism spectrum disorders: a multidimensional approach. Sleep. 2006 Dec;29(12):1563-71. doi: 10.1093/sleep/29.12.1563. PMID 17252887
- [Background] Richdale AL, Schreck KA. Sleep problems in autism spectrum disorders: prevalence, nature, & possible biopsychosocial aetiologies. Sleep Med Rev. 2009 Dec;13(6):403-11. doi: 10.1016/j.smrv.2009.02.003. Epub 2009 Apr 24. PMID 19398354
- [Background] Taylor MA, Schreck KA, Mulick JA. Sleep disruption as a correlate to cognitive and adaptive behavior problems in autism spectrum disorders. Res Dev Disabil. 2012 Sep-Oct;33(5):1408-17. doi: 10.1016/j.ridd.2012.03.013. Epub 2012 Apr 21. PMID 22522199
- [Background] Wasdell MB, Jan JE, Bomben MM, Freeman RD, Rietveld WJ, Tai J, Hamilton D, Weiss MD. A randomized, placebo-controlled trial of controlled release melatonin treatment of delayed sleep phase syndrome and impaired sleep maintenance in children with neurodevelopmental disabilities. J Pineal Res. 2008 Jan;44(1):57-64. doi: 10.1111/j.1600-079X.2007.00528.x. PMID 18078449

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Most patients were recruited from the clinical practice of the Principal Investigator. We also posted flyers in the hospital outpatient clinics and sent "Dear Physician" recruitment letters to other pediatric neurologists and psychologists in our catchment area.
Groups:
- Group A: Group A received an initial 5 week Run-In Period where other medications were withdrawn, and Placebo medication was given. Instructions for improving sleep hygiene were given during this phase.
  This Run-In Period was followed by Phase 1 (5 weeks) with active study medication (donepezil and melatonin) with dose based on subject age/weight.
  This was followed by Phase 2 (5 weeks) with continued study medication. At the conclusion of Phase 2, study medication was discontinued and a variable washout period (2-12 weeks) followed, ending with the next scheduled clinic visit with the Principal Investigator.
- Group B: Group B received an initial 5 week Run-In Period where other medications were withdrawn, and Placebo medication was given. Instructions for improving sleep hygiene were given during this phase.
  This Run-In Period was followed by Phase 1 (5 weeks)where Placebo medication was continued.
  This was followed by Phase 2 (5 weeks) with active study medication (donepezil and melatonin) with dose based on subject age/weight.
  At the conclusion of Phase 2, study medication was discontinued and a variable washout period (2-12 weeks) followed, ending with the next scheduled clinic visit with the Principal Investigator.
Period: Run-In Phase (5 Weeks)
Arm/Group | Group A | Group B
Started | 4 | 8
Completed | 3 | 6
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2
Period: Phase 1 (5 Weeks)
Arm/Group | Group A | Group B
Started | 3 | 6
Completed | 2 | 6
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Phase 2 (5 Weeks)
Arm/Group | Group A | Group B
Started | 2 | 6
Completed | 2 | 6
Not Completed | 0 | 0
Period: Wash-Out Phase (2-12 Weeks)
Arm/Group | Group A | Group B
Started | 2 | 6
Completed | 2 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group A; Group B: Melatonin and donepezil (melatonin 3mg and donepezil 1.25-5mg based on age/weight each night) or placebo for 15 weeks
  Melatonin and Donepezil: The duration depends on group assignment.
  Placebo: The duration depends on group assignment.
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 4 | 8 | 12
Age, Continuous [Median (Full Range); unit: years] | 11 [7 to 15] | 9.5 [7 to 16] | 9.5 [7 to 16]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 4 | 7 | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 4 | 8 | 12
ABC Lethargy/Social Withdrawal [Median (Full Range); unit: units on a scale] — Subscale of the Aberrant Behavior Checklist (ABC). The checklist is widely used in research with children with autism. It is considered sensitive to drug effects. The Lethargy/Social Withdrawal subscale contains items such as: "Listless, sluggish, inactive" ; "Withdrawn, prefers solitary activities"; "Does not try to communicate by words or gestures"; "Shows few social reactions to others". The subscale consists of 16 items, each rated on a 4 point scale (0 = not at all, 3 = severe). Possible scores range from 0 to 48. Higher scores mean more lethargy and/or more social withdrawal.
  units on a scale | 8 [3 to 23] | 10 [5 to 28] | 9.5 [3 to 28]
ABC Stereotypic Behavior [Median (Full Range); unit: units on a scale] — Subscale of the ABC Checklist, which is considered sensitive to drug effects. The Stereotypic Behavior subscale contains items such as: "Meaningless, recurring body movements" ; "Odd, bizarre in behavior"; "Waves, shakes the extremities repeatedly"; "Rocks body back and forth".
  The subscale consists of 7 items, each rated on a 4 point scale (0 = not at all, 3 = severe). Possible scores range from 0 to 21. Higher scores mean more stereotyped behavior.
  units on a scale | 7.5 [3 to 12] | 7.5 [1 to 15] | 7.5 [1 to 15]
Sleep Duration (hours) [Median (Full Range); unit: hours] — As measured by the Child's Sleep Habits Questionnaire (CSHQ).
  hours | 8.2 [7 to 9] | 7 [4.5 to 8] | 7.1 [4.5 to 9]

OUTCOME MEASURES:

1. Primary Outcome: Aberrant Behavior Checklist (ABC) Lethargy/Social Withdrawal Subscale
Description: Subscale of the Aberrant Behavior Checklist (ABC). Subscales were derived by factor analysis (n=927).
  The checklist was first developed for use with severely mentally retarded individuals. More recently it has become widely used in research with children with autism. The ABC checklist is considered sensitive to drug effects.
  The Lethargy/Social Withdrawal subscale contains items such as: "Listless, sluggish, inactive" ; "Withdrawn, prefers solitary activities"; "Does not try to communicate by words or gestures"; "Shows few social reactions to others".
  The subscale consists of 16 items, each rated on a 4 point scale (0 = not at all, 3 = severe). Possible scores range from 0 to 48. Higher scores mean more lethargy and/or more social withdrawal.
Time Frame: Subscale rating was made by parent/caregiver every 5 weeks for a total of 5 times. Due to small N, only the endpoint of the study is reported here. Study endpoint (Visit 5) was after at least 18 wks, including 2 wks of washout, up to a maximum of 27 wks.
Population: Participants who completed the trial.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Group A | Group B
Number analyzed (Participants) | 2 | 6
score on a scale | 6 [0 to 12] | 5.5 [1 to 33]

2. Secondary Outcome: Aberrant Behavior Checklist (ABC) Stereotypic Behavior Subscale.
Description: Subscale of the Aberrant Behavior Checklist (ABC). Subscales were derived by factor analysis (n=927).
  The checklist was first developed for use with severely mentally retarded individuals. More recently it has become widely used in research with children with autism. The ABC Checklist is considered sensitive to drug effects.
  The Stereotypic Behavior subscale contains items such as: "Meaningless, recurring body movements" ; "Odd, bizarre in behavior"; "Waves, shakes the extremities repeatedly"; "Rocks body back and forth".
  The subscale consists of 7 items, each rated on a 4 point scale (0 = not at all, 3 = severe). Possible scores range from 0 to 21. Higher scores mean more stereotyped behavior.
Time Frame: as for outcome 1
Population: Participants who completed the trial.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Group A | Group B
Number analyzed (Participants) | 2 | 6
score on a scale | 6 [4 to 8] | 2.5 [1 to 11]

3. Secondary Outcome: Sleep Duration (Hours)
Description: A brief seven item questionnaire adapted from the Children's Sleep Habits Questionnaire (CSHQ). This parental questionnaire assesses sleep behaviors in children. It has been validated in children with ASD, correlates with polysomnographic recordings, and has been used successfully in previous studies of melatonin with such children. The CSHQ items chosen for this study come from the subscales found to be most often disturbed in children with autism.
Time Frame: Rating was made by parent/caregiver every 5 weeks for a total of 5 times. Due to small N, only the endpoint of the study is reported here. Study endpoint (Visit 5) was after at least 18 wks, including 2 wks of washout, up to a maximum of 27 wks.
Population: Participants who completed the trial.
Measure: Median (Full Range); unit: hours
Arm/Group | Group A | Group B
Number analyzed (Participants) | 2 | 6
hours | 8.75 [8 to 9.5] | 6.9 [5 to 10]

4. Secondary Outcome: Clinical Global Impressions Scale, Clinician Impression of Global Improvement
Description: Measured by the Clinical Global Impressions Scale. The Clinician Impression of Global Improvement is a single item rated as follows:
  1 = very much improved; 2 = much improved; 3 = minimally improved; 4 = no change; 5 = minimally worse; 6 = much worse; 7 = very much worse. Thus, higher scores indicate a change for the worse. Note: This measure was not evaluated at Baseline.
Time Frame: Rating was made by clinician every 5 weeks for a total of 5 times. Due to small N, only the endpoint of the study is reported here. Study endpoint (Visit 5) was after at least 18 wks, including 2 wks of washout, up to a maximum of 27 wks.
Population: Participants who completed the trial.
Measure: Median (Full Range); unit: units on a scale, where 4=no change
Arm/Group | Group A | Group B
Number analyzed (Participants) | 2 | 6
units on a scale, where 4=no change | 3 [3 to 3] | 5 [2 to 6]

5. Secondary Outcome: Clinical Global Impressions Scale, Parent Reported Global Improvement
Description: Parent Impression of Global Improvement is a single item rated as follows:
  1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; 7=very much worse. Thus, higher scores indicate a change for the worse. Note: This measure was not evaluated at Baseline.
Time Frame: Rating was made by parent every 5 weeks for a total of 5 times. Due to small N, only the endpoint of the study is reported here. Study endpoint (Visit 5) was after at least 18 wks, including 2 wks of washout, up to a maximum of 27 wks.
Population: Participants who completed the trial.
Measure: Median (Full Range); unit: units on a scale, where 4=no change
Arm/Group | Group A | Group B
Number analyzed (Participants) | 2 | 6
units on a scale, where 4=no change | 2.8 [2 to 3.5] | 3.5 [2 to 5]

ADVERSE EVENTS:
Time Frame: Overall study - Baseline thru Visit 4, a maximum of 27 weeks. This includes a 5 week run-in period with Placebo, 10 weeks of active study drug (Group A) vs. an additional 5 weeks of placebo followed by 5 weeks of active study drug (Group B), and 2-12 weeks of follow-up, ending with the next scheduled clinic visit with the Principal Investigator. There was no post-study follow-up.
Description: The parent/guardian was queried about adverse events at each study visit. These events were discussed with the Principal Investigator and the study coordinator.
Arm/Group | Group A | Group B
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/8
Other Adverse Events (participants affected / at risk) | 2/4 | 2/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (N=4) | Group B (N=8)
difficulty falling asleep (Nervous system disorders) | 2 | 2

LIMITATIONS AND CAVEATS:
No statistical comparisons were undertaken due to the small sample size in the two groups. Study enrollment/completion proved insufficient to permit any conclusions to be drawn. Enrollment/completion was likely limited because of the study requirement that all prior sleep medications, including melatonin, be discontinued as a condition for study participation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-23): https://cdn.clinicaltrials.gov/large-docs/82/NCT02487082/Prot_SAP_000.pdf